CLINICAL TRIAL: NCT04291235
Title: The NEUROlogically-impaired Extubation Timing Trial
Brief Title: The NEUROlogically-impaired Extubation Timing Trial (NEURO-ETT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Damon Scales, Chief of Critical Care Medicine, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NEURO-ETT
Record Dates: First submitted 2020-02-03; First posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Acute Brain Injury
Keywords: Subarachnoid Hemorrhage; Diffuse Axonal Injury; Ischemic Stroke; Intracerebral Hemorrhage; Brain Tumor; Global Cerebral Anoxia/Cardiac Arrest; Meningitis/Encephalitis; Cerebral Abscess; Epidural Hematoma; Subdural Hematoma; Seizure
MeSH Terms: conditions — Brain Injuries; Subarachnoid Hemorrhage; Diffuse Axonal Injury; Ischemic Stroke; Cerebral Hemorrhage; Brain Neoplasms; Heart Arrest; Meningitis; Encephalitis; Brain Abscess; Hematoma, Epidural, Spinal; Hematoma, Subdural; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Airway Management Pathway (Active Comparator): An airway management pathway consisting of daily assessments and removal of the breathing tube as soon as patients can breathe on their own and appear able to protect their airway
  Interventions: Procedure: Airway Management Pathway
- Usual Care (Active Comparator): The usual clinical practice is often to keep the patient on artificial respiration for longer in the hope that the patient will wake up before removing the tube, or performing a tracheostomy if the patient doesn't wake up
  Interventions: Procedure: Usual Care

INTERVENTIONS:
Procedure: Airway Management Pathway — Patients in this group will receive several components that comprise airway management pathway: (1) daily spontaneous breathing trials (SBTs); (2) prompt extubation following successful extubation readiness criteria; (3) high-flow nasal oxygen for at least 24 hours following extubation.
  Arms: Airway Management Pathway
Procedure: Usual Care — Patients in this group will be treated according to usual care, which may include extubation or tracheostomy timed according to treating physicians' discretion.
  Arms: Usual Care

SUMMARY:
This trial in brain-injured patients will test which of the following will lead to better patient outcomes: (1) an airway management pathway consisting of daily assessments and removal of the breathing tube as soon as patients can breathe on their own and appear able to protect their airway; versus (2) the usual treatment patients would have received if they were not enrolled in this trial.

DETAILED DESCRIPTION:
Thousands of patients suffer severe brain injuries every year, from causes such as trauma, stroke, and infection. These patients are usually not fully awake and need help with their breathing and with preventing them from choking on their secretions. This is done with a breathing tube inserted through the mouth into the lungs and connected to a breathing machine. As patients recover, It is often unclear when the best time is to remove the breathing tube. Doctors might decide to remove it relatively early, or they may wait until the patient is more fully awake, or they may perform a tracheostomy (neck surgery to insert a new tube directly into the windpipe (trachea), replacing the temporary breathing tube). Each of these approaches has risks and benefits. This trial in brain-injured patients will test which of the following will lead to better patient outcomes: (1) an airway management pathway consisting of daily assessments and removal of the breathing tube as soon as patients can breathe on their own and appear able to protect their airway; versus (2) the usual treatment patients would have received if they were not enrolled in this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 16 years
2. Acute brain injury (subarachnoid hemorrhage, diffuse axonal injury, ischemic stroke, intracerebral hemorrhage, brain tumor, global cerebral anoxia/cardiac arrest, meningitis/encephalitis, cerebral abscess, epidural hematoma, subdural hematoma, seizure) that occurred within the previous 4 weeks
3. Receiving mechanical ventilation via endotracheal tube for ≥ 48 hours

Exclusion Criteria:

1. Quadriplegic
2. Neuromuscular disease that will result in prolong need for mechanical ventilation, including but not limited to Guillain-Barre syndrome, cervical spinal cord injury, advanced multiple sclerosis
3. Do-Not-Reintubate order in place
4. Previously randomized in this trial
5. Underlying pre-existing condition with life expectancy less than 6-months
6. Current enrolment in an RCT that precludes NEURO-ETT co-enrollment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Total Duration of Mechanical Ventilation | Up to 60 Days
  Total duration of mechanical ventilation (to 60 days) accounting for the competing risk of death

SECONDARY OUTCOMES:
Mortality at ICU discharge and Hospital Discharge | ICU Discharge, Hospital Discharge, 3 months, and 6 months
  Mortality at ICU Discharge, Hospital Discharge, 3 months, and 6 months
Ventilator-Free Days at Day 60 | Up to 60 days
  Days alive and not receiving mechanical ventilation
ICU Free Days At Day 60 | Up to 60 Days
  ICU free days (days alive and not spent in an ICU)
Airway or Tracheostomy complications | Up to 30 days
  Presence versus absence of airway complication
Nutrition Intake | Up to 6 Months
  Time to normal oral nutrition intake
Antibiotics Days | Up to 30 Days
  Injection or infusion of antibiotics given intravenously
Tracheostomy Rates | Up to 6 Months
  Presence versus absence of tracheostomy insertion
ICU Readmission Rates | Hospital discharge, up to 90 days
  ICU readmission rates to hospital discharge
Discharge Destination | Hospital discharge, up to 90 days
  Discharge destination for the patient post hospitalization
Extended Glasgow Outcome Score | 3 months and 6 months
  Minimum score 1 (worst) to maximum score 8 (best) at 3 months and 6 months
EuroQol-5D | 3 months and 6 months
  Minimum score 1 (worst) to maximum score 100 (best) at 3 months and 6 months
Delirium Free Days | Up to 30 Days
  Days alive and free of delirium while in ICU up to day 30

CONTACTS AND LOCATIONS:
Overall Officials: Niall Ferguson, MD, MSc, Principal Investigator — Toronto General Hospital; Damon Scales, MD, PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (14):
- Canada (14):
  - University of Alberta Hospital, Edmonton, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Hamilton General Hospital, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec
  - L'Hôpital de l'Enfant-Jésus, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Angriman F, Amaral ACKB, Fan E, Taran S, McCredie VA, Baker A, Bosma KJ, Brochard LJ, Adhikari NKJ, Cuthbertson BH, Scales DC, Ferguson ND. Timing of Extubation in Adult Patients with Acute Brain Injury. Am J Respir Crit Care Med. 2025 Mar;211(3):339-346. doi: 10.1164/rccm.202408-1553OC. PMID 39585965